CLINICAL TRIAL: NCT04733235
Title: The Effect of Progesterone Induced Endometrial Compaction on Pregnancy Outcomes in Frozen-thawed Embryo Transfer at the Blastocyst Stage
Brief Title: the Effect of Endometrial Compaction Caused by Progesterone Effect on Pregnancy Outcomes
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, ŞAFAK OLGAN, ASSOCIATE PROFESSOR, Akdeniz University
Other Study IDs: AkdenizUKD
Record Dates: First submitted 2021-01-17; First posted 2021-02-02 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Infertility; Female Infertility; Frozen-thawed Embryo Transfer
Keywords: infertility; female infertility; frozen- thawed embryo transfer; female
MeSH Terms: conditions — Infertility; Infertility, Female | interventions — Progesterone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with endometrial compaction: Participants who have endometrial compaction caused by progesterone effects on undergoing frozen embryo transfer with artificial hormone replacement
  Interventions: Drug: Progesterone
- without endometrial compaction: Participants who have not endometrial compaction caused by progesterone effects on undergoing frozen embryo transfer with artificial hormone replacement
  Interventions: Drug: Progesterone

INTERVENTIONS:
Drug: Progesterone — ultrasound measurements of endometrial thickness at the end of the estrogen phase and the day of embryo transfer.
  Other Names: Diagnostic Test: Blood test Measurement of E2, P4, LH, FSH hormones Diagnostic Test: Transvaginal

SUMMARY:
The purpose of this prospective cohort study is to assess the effect of endometrial compaction caused by progesterone effect on pregnancy outcomes

DETAILED DESCRIPTION:
For a pregnancy to occur, the embryo must implant in a receptive endometrium during the window of implantation, which is thought to occur from day 22 to 24 of an idealized 28-day cycle. Early studies have suggested that assessing endometrial thickness with the use of ultrasound may be an alternative to invasive techniques such as endometrial biopsy for attempting to determine a receptive endometrium for frozen-thawed embryo transfer (FET).

A preovulatory endometrial thickness of 7 mm or more is considered to be the cutoff for endometrial receptivity, below which many physicians would cancel an embryo transfer. However, in most studies in the literature, endometrial thickness was measured either on the day of hCG in fresh embryo transfer cases or on the last day of estrogen treatment in thawed embryo transfers. There are a limited number of studies evaluating the luteal period, embryo transfer day and endometrial thickness.

Accordingly, in this prospective cohort study is to assess the effect of endometrial compaction caused by progesterone effect on pregnancy outcomes

ELIGIBILITY:
Inclusion Criteria:

1. Woman aged 18-40 years
2. Presence of high quality (>2BB) blastocyst
3. Hormonal(estrogen and progesterone) frozen- thawed embryo transfer cycles
4. presence of high quality blastocyst cryopreserved by vitrification method.
5. A single embryo transfer

Exclusion Criteria:

1. Presence of uterine pathology
2. Participants whose optimal endometrial image cannot be obtained due to uterine position
3. Participants whose treatments were canceled for any reason before embryo transfer
4. Participants which had embryo transfer on the day 2 or 3 (at the cleavage stage)
5. Participants who had 2 embryo transfer
6. Presence of low quality (<2BB) blastocyst
7. > 15% loss of viability in the embryo during embryo thawing

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female patients underwent infertility treatment
Study Population: Women underwent frozen embryo transfer
Sampling Method: Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
The change in endometrial thickness | 1 year
  changing in millimeters of endometrial thickness at the end of the estrogen phase and the day of embryo transfer.
ongoing pregnancy rates. | 1 year
  pregnancy beyond 12 weeks of gestational age.

SECONDARY OUTCOMES:
The Correlation of Serum Progesterone Levels With the Degree of Endometrial Compaction on the Day of Frozen Embryo Transfer | On the day of frozen embryo transfer
  comparison of progesterone levels and endometrial thickness
Clinical pregnancy rate | 6-7 weeks after the last menstrual period of the patient
  6th week gestational age
Implantation rate | 5 weeks after the last menstrual period of the patient
  Percentage of gestational sacs compared to the number of embryos transferred
Clinical miscarriage | after 5th gestational week
  pregnancy loss after ultrasonographic detection of an intrauterine gestational sac

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Haas J, Smith R, Zilberberg E, Nayot D, Meriano J, Barzilay E, Casper RF. Endometrial compaction (decreased thickness) in response to progesterone results in optimal pregnancy outcome in frozen-thawed embryo transfers. Fertil Steril. 2019 Sep;112(3):503-509.e1. doi: 10.1016/j.fertnstert.2019.05.001. Epub 2019 Jun 24. PMID 31248618